CLINICAL TRIAL: NCT02763423
Title: The Efficacy of Allogeneic Umbilical Cord Mesenchymal Stem Cell Transplantation to Treat New-onset Type 1 Diabetes With Diabetic Ketoacidosis
Brief Title: Allogeneic Umbilical Cord Mesenchymal Stem Cell Transplantation for Type 1 Diabetes With Diabetic Ketoacidosis
Acronym: UCMSCDKA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Dalong Zhu, Chief Physician, Professor, Director of Endocrinology Department, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJGYNFM-SC-02
Record Dates: First submitted 2016-04-19; First posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Ketoacidosis, Diabetic
Keywords: umbilical cord stem cell; diabetic ketoacidosis
MeSH Terms: conditions — Diabetic Ketoacidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- umbilical cord mesenchymal stem cell (Experimental): single- or double-dose intravenous injection of umbilical cord mesenchymal stem cells for the treatment of severe type 1 diabetes patients
  Interventions: Procedure: umbilical cord mesenchymal stem cell

INTERVENTIONS:
Procedure: umbilical cord mesenchymal stem cell — allogeneic umbilical cord mesenchymal stem cell transplantation by intravenous injection

SUMMARY:
This is a phase II trial in individuals who have been diagnosed with type 1 diabetes within the previous 12 months and suffered from diabetic ketoacidosis at onset of disease. The purpose of this study is to determine whether allogeneic umbilical cord mesenchymal stem cell transplantation is effective in the treatment of patients with severe type 1 diabetes.

DETAILED DESCRIPTION:
To assess the clinical efficacy of allogeneic umbilical cord mesenchymal stem cell transplantation in the treatment of patients with severe type 1 diabetes, defined as with the history of diabetic ketoacidosis from diagnosis. All the patients are intravenously administrated with single-dose or double-dose umbilical cord mesenchymal stem cell and followed up for 36 months. Clinical and laboratory manifestations are compared before and after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Duration of disease less than 12 months from diagnosis
* With the history of diabetic ketoacidosis

Exclusion Criteria:

* Pregnancy
* Severe psychiatric disorder
* Severe organic impairment(renal,hepatic,cardiac,pulmonary)
* Active infectious disease
* Previous or present neoplastic disease

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline exogenous insulin dose at different time points post treatment | 1 month, 3 months,6 months, 12 months, 24 months, 36 months

SECONDARY OUTCOMES:
C-peptide level | 1 month, 3 months, 6 months, 12 months, 24 months, 36 months
HbA1c level | 1 month, 3 months, 6 months, 12 months, 24 months, 36 months
titres of islet antigen antibodies | 1 month, 3 months, 6 months, 12 months,24 months, 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Zhu, MD.PhD., Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- The affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang W, Ling Q, Wang B, Wang K, Pang J, Lu J, Bi Y, Zhu D. Comparison of therapeutic effects of mesenchymal stem cells from umbilical cord and bone marrow in the treatment of type 1 diabetes. Stem Cell Res Ther. 2022 Aug 8;13(1):406. doi: 10.1186/s13287-022-02974-1. PMID 35941696